CLINICAL TRIAL: NCT06726577
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial Evaluating the Safety, Efficacy, and Pharmacokinetic Characteristics of TP04HN106 in the Treatment of Patients With Amyotrophic Lateral Sclerosis
Brief Title: TP04HN106 in the Treatment of Patients With Amyotrophic Lateral Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Talengen Institute of Life Sciences, Shenzhen, P.R. China. (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TP04HN106-ALS-IIT
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental drug group (Experimental)
  Interventions: Drug: TP04HN106
- Placebo group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: TP04HN106 — During the treatment period, the experimental drug group received intravenous injections of 0.83mL/kg TP04HN106 each time; During the extension period, all subjects received intravenous injection of 0.83mL/kg TP04HN106.
  Arms: Experimental drug group
Drug: Saline — The placebo group received intravenous injections of 0.83mL/kg of saline each time. In the experiment, all subjects received Liraglutide tablets as the standard baseline treatment.
  Arms: Placebo group

SUMMARY:
This trial adopts a multicenter, randomized, double-blind, placebo-controlled parallel design.

This experiment is divided into two groups: the experimental drug group and the placebo group. Successful participants will be randomly assigned to the two groups, with an expected enrollment of 60 participants. There will be 30 participants in the experimental drug group and 30 participants in the placebo group. During the treatment period, the experimental drug group received intravenous injections of 0.83mL/kg TP04HN106 each time; The placebo group received intravenous injections of 0.83mL/kg of saline each time. During the extension period, all subjects received intravenous injection of 0.83mL/kg TP04HN106. In the experiment, all subjects received Liraglutide tablets as the standard baseline treatment.

The subjects who were successfully screened in the experiment were enrolled in sequence, and the safety, tolerability, efficacy, and pharmacokinetic characteristics of the experimental drug were evaluated after administration. The entire trial includes a screening period of 1 week, a treatment period of 12 weeks (including 3 treatment cycles, each treatment cycle of 4 weeks), an extension period of 12 weeks (including 3 treatment cycles, each treatment cycle of 4 weeks), and a follow-up period of 4 weeks. In addition, some subjects underwent a 1-week single dose PK study before the start of the treatment period; In addition, during the first treatment cycle of the treatment period, some subjects were selected for multiple dosing PK studies.

We plan to conduct a single dose PK study among 12 subjects, with 6 subjects in the experimental group and 6 subjects in the control group; Multiple dose PK studies were conducted among 12 subjects, with 6 subjects in the experimental group and 6 sujects in the control group. It is not allowed for the same subject to participate in both single dose and multiple dose PK studies simultaneously.

The 1st to 12th subjects planned to be enrolled in the trial will undergo a single dose PK study. After the first dose, venous blood will be collected from the 12 subjects according to the blood sample collection requirements, and their PK characteristics will be evaluated. The observation period for single dose administration is one week. After completing the final blood sample collection and safety assessment, the subjects enter the treatment period, extension period, and follow-up period.

The 13th to 24th subjects planned to be enrolled in the trial will undergo multiple dose PK studies. These 12 subjects will have their venous blood collected according to the blood sample collection requirements during the first treatment cycle of the treatment period, and their PK characteristics will be evaluated. After completing the treatment period, the subjects will enter the extension period and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for amyotrophic lateral sclerosis (ALS) (Gold Coast Criteria 2020）;
2. Age ≥18 years old, male or female;
3. The amyotrophic lateral sclerosis Function Rating Scale (ALSFRS-R）of pre-visit subjects should be ≥1 score for dyspnea, upright breathing and respiratory dysfunction;
4. Pre-randomized subjects received stable dose of riluzole tablets for ≥7 days, and should maintain the treatment until the last study visit;
5. Voluntarily participate in clinical trials, sign informed consent, and understand and comply with study procedures.

Exclusion Criteria:

1. The subject is known to be allergic to the investigational drug or its excipients;
2. The subject has a disease or injury that interferes with functional assessment or threatens life, or is accompanied by a serious irreversible disease of the heart, lung, liver, or brain, or is accompanied by a failure of different organs (for patients with respiratory failure, only patients diagnosed as type I or type II respiratory failure are excluded);
3. The subject has a major mental illness or cognitive dysfunction;
4. Patients with a history of secondary or above surgery within one month before the screening period;
5. The subjects participated in other clinical studies within 1 month;
6. The subjects are pregnant or lactating women;
7. Poor compliance or other researchers believe that there are any circumstances that are not suitable for inclusion.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Rating Scale (ALSFRS-R) | Baseline, 10th week
  The Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) measures the severity of functional disorders. This scale measures three functional domains, namely medullary function, motor function, and respiratory function. The evaluation will consist of 12 questions, with scores ranging from 0 (non functional) to 4 (fully functional), for a total score of 48, which will indicate the highest level of functionality.

SECONDARY OUTCOMES:
ALSFRS-R | Baseline, week 2, 6, 12, 14, 18, 22, and 28
  The Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) measures the severity of functional disorders. This scale measures three functional domains, namely medullary function, motor function, and respiratory function. The evaluation will consist of 12 questions, with scores ranging from 0 (non functional) to 4 (fully functional), for a total score of 48, which will indicate the highest level of functionality.
Rasch Global Disability Assessment Scale (ROADS) scores | Baseline, week 2, 6, 10, 12, 14, 18, 22, and 28
  The Rasch Global Disability Assessment Scale (ROADS) scores is a comprehensive functional impairment assessment scale for amyotrophic lateral sclerosis syndrome. This scale consists of 28 items, arranged in order from the easiest action to the most difficult action, with a total score of 56 points
FVC% | Basline, week 6, 10, 12, 14, 18, 22, and 28
  The change value/rate of FVC% compared to baseline at weeks 6, 10, 12, 14, 18, 22, and 28;
Muscle strength | Baseline，week 2, 6, 10, 12, 14, 18, 22, and 28;weeks 2, 6, 10, 12, 14, 18, 22, and 28
  Changes in muscle strength from baseline as measured by a handheld dynamometer (HHD) at weeks 2, 6, 10, 12, 14, 18, 22, and 28;
Neurofilament light chain level | Baseline，week 10，week 22
  Change in the levels of Neurofilament light chain (NFL) in the subjects' venous plasma at week 10 and 22
CMAP amplitude | Baseline，week 10，week 22
  Changes in neuromuscular electrophysiological examination (CMAP amplitude measurement of clinically affected area) relative to baseline at week 10 and 22.
Incidence of permanent invasive breathing or oxygen assistance/death | Through study completion, an average of 28 weeks
  Incidence of permanent invasive breathing or oxygen assistance/death during the trial;

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China